CLINICAL TRIAL: NCT04463784
Title: Peking Union Medical College Hospital
Brief Title: Efficacy of Efavirenz 400mg vs. 600mg Combined With Lamivudine and Tenofovir in Treatment Naive HIV Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LI Taisheng, Chief, Department of Infectious Diseases, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CACT 1809
Record Dates: First submitted 2018-07-15; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: HIV/AIDS; Mental Impairment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — efavirenz; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efavirenz 400MG Oral Tablet (Experimental): Recruited treatment-naive HIV infected patients will be given Lamivudin 300mg per day, tenofovir 300mg per day and efavirenz 400mg per day as antiretroviral treatment.
  Interventions: Drug: Efavirenz 400Mg Oral Tablet
- Efavirenz 600MG Oral Tablet (Active Comparator): Recruited treatment-naive HIV infected patients will be given Lamivudin 300mg per day, tenofovir 300mg per day and efavirenz 600mg per day, per standard dose.
  Interventions: Drug: Efavirenz 600Mg Oral Tablet

INTERVENTIONS:
Drug: Efavirenz 400Mg Oral Tablet — The experimental arm will receive 400mg efavirenz per randomization with other two antiretroviral medication (tenofovir and lamivudine).
  Arms: Efavirenz 400MG Oral Tablet
Drug: Efavirenz 600Mg Oral Tablet — The active comparator arm will receive 600mg efavirenz per randomization with other two antiretroviral medication (tenofovir and lamivudine).
  Arms: Efavirenz 600MG Oral Tablet

SUMMARY:
The present study will be a randomized controlled study in which 500 treatment-naive HIV patients will be randomized 1:1 to Efaviren 400mg v.s. 600mg combined with lamivudine and tenofovir. The whole cohort will be followed for two years. Efficacy and safety of each regimen will be evaluated throughout the study.

DETAILED DESCRIPTION:
As efaviren has been commonly used as the first-line therapy in HIV infection worldwide, its major side effect i.e. the mental effects have been noticed and has a major influence on the adherence and efficacy of ART regimen. Mental effects of efaviren have been especially critical in Chinese patients, as the effective and toxic ranges of efaviren plasma concentration in Chinese patients are very close to each other.

In this study, 500 treatment-naive Chinese patients with a body weight < 60kg will be screened and recruited. Patients will be randomized 1:1 to efaviren 400mg v.s. 600mg combined with lamivudine and tenofovir. All patients will be followed regularly for 2 years, at 0, 2w, 4w, 3m and every 3 months. Virological and immunological measurements will be done at each visit. Meanwhile, various mental scales will be performed at each visit to evaluate the mental effects of each arm.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Willingness and availability to engage in study activities for the duration of the study
* Age between 18-65
* Documented HIV-1 infection (confirmed by Western blot)
* Received no prior antiretroviral therapy

Exclusion Criteria:

* Pregnancy or breastfeeding or anticipated pregnancy in two years
* History of AIDS-defining illness
* Hemoglobin < 9g/dl；or peripheral white blood cell counts < 2000/μl；or neutrophil counts < 1000 /μl；or platelet count < 75,000/μl；
* Liver disease (transaminase and alkaline phosphatase levels more than three times the upper limit of the normal range (ULN), bilirubin level more than 2.5 times the ULN)
* Chronic kidney disease (serum creatinine level more than 1.5 times the ULN)
* Patients with a history of injection drug usage
* Patients with a history of mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Virological measurements at 12 weeks | 12 weeks
  Plasma viral load
Change from Baseline Virological measurements at 24 weeks | 24 weeks
  Plasma viral load
Change from Baseline Virological measurements at 48 weeks | 48 weeks
  Plasma viral load
Change from Baseline Virological measurements at 72 weeks | 72 weeks
  Plasma viral load
Change from Baseline Virological measurements at 96 weeks | 96 weeks
  Plasma viral load
Change from Baseline Immunological measurements at 12 weeks | 12 weeks
  CD4 T cell count
Change from Baseline Immunological measurements at 24 weeks | 24 weeks
  CD4 T cell count
Change from Baseline Immunological measurements at 48 weeks | 48 weeks
  CD4 T cell count
Change from Baseline Immunological measurements at 72 weeks | 72 weeks
  CD4 T cell count
Change from Baseline Immunological measurements at 96 weeks | 96 weeks
  CD4 T cell count

SECONDARY OUTCOMES:
Adverse effects measured by Dizziness Handicap Inventory | 0, 12, 24, 48, 72, 96 weeks
  Measure statistically significant difference in perception of dizziness by administering the Dizziness Handicap Inventory (DHI) between two groups at different time point. The 25-item tool comprises three sub-scales: physical (DHI-P; 7 items), emotional (DHI-E; 9 items), and functional (DHI-F; 9 items) and each item is scored from 0 to 4. Grading standard: 0-30 points is defiend as minor obstacles, 31-60 points as moderate obstacle, and 61-100 points as serious obstacle with high risk of falling.
Adverse effects measured by Hamilton Depression Scale-24 | 0, 12, 24, 48, 72, 96 weeks
  Measure statistically significant difference in perception of depression by administering the Hamilton Depression Scale-24 (HAMD-24) between two groups at different time point. The Hamilton Depression Rating Scale (HAMD) has a total of 24 items. 14 items were scored from 0 to 4, and 10 items were scored from 0 to 2. The total score that less than 8 points is defined as no depression, 8 to 20 points as may be depression, scores that more than 20 is defined as mild or moderate depression, and more than 35 points as severe depression.
Adverse effects measured by Pittsburgh Sleep Quality Index | 0, 12, 24, 48, 72, 96 weeks
  Measure statistically significant difference in perception of sleep quality by administering the Pittsburgh Sleep Quality Index (PSQI) between two groups at different time point. PSQI was used to assess the sleep quality of subjects in the last month. It consists of 19 self-evaluation items and 5 other evaluation items, of which only 18 self-evaluation items participate in scoring. 18 items constitute 7 components, and each component is scored according to 0 ~ 3 grades. The PSQI total score ranges from 0 to 21. The higher the score indicates the worser sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, PhD, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tongtong Y, Shenghua H, Yin W, Lin C, Huanxia L, Chunrong L, Ruifeng Z, Xiaojing Y, Yuan Y, Yuanhong H, Ke Y. Effectiveness and Safety of Dolutegravir Versus Efavirenz-Based Antiviral Regimen in People Living With HIV-1 in Sichuan Province of China: A Real-World Study. J Acquir Immune Defic Syndr. 2022 Oct 1;91(S1):S1-S7. doi: 10.1097/QAI.0000000000003041. PMID 36094508